CLINICAL TRIAL: NCT02421302
Title: The Role of Nutrition as a Determinant of Immune Function and Pharmacological Outcome Amongst HIV Infected Malnourished Children in Uganda
Brief Title: The Pediatric HIV Nutrition Study in Uganda
Acronym: NOURISH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Infectious Diseases Institute (Other)
Collaborators: University of Dublin, Trinity College (Other)
Responsible Party: Sponsor-Investigator, Infectious Diseases Institute, PhD Candidate, Makerere University
Organization: Makerere University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ST/0110/15; ST/0110/15 (Registry Identifier: Nutrition Study Pead.)
Record Dates: First submitted 2015-02-18; First posted 2015-04-20 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Child Nutrition Disorders
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Well-nourished HIV+ ART naive (No Intervention): These children aged between 6months-12years will be followed up for 12weeks to look at their nutrition, immune and pharmacological responses. They will receive routine nutritional and ART adherence counseling
- Moderately-malnourished HIV+; RUTF (Active Comparator): These children aged between 6months - 12years, ART naive or experienced, will be initiating ready-to-use-therapeutic(RUTF) food and will be followed up for 12 weeks to see the effect of nutrition supplementation on immune and pharmacological responses
  Interventions: Dietary Supplement: RUTF
- Severely acute-malnourished HIV+; RUTF (Active Comparator): These children aged between 6months - 12years, ART naive or experienced, will be initiating ready-to-use-therapeutic(RUTF) food and will be followed up for 12 weeks to see the effect of nutrition supplementation on immune and pharmacological responses
  Interventions: Dietary Supplement: RUTF

INTERVENTIONS:
Dietary Supplement: RUTF — This is ready-to-use-therapeutic-food
  Other Names: Ready-to-Use-Therapeutic-Food
  Arms: Moderately-malnourished HIV+; RUTF; Severely acute-malnourished HIV+; RUTF

SUMMARY:
This will be cohort study design with both qualitative and quantitative methods of data collection. The investigators are aiming to study 64 HIV positive children as healthy controls either initiating ART or already on ART and 86 malnourished HIV infected children on ART or naïve initiating ART and RUTF aged between 6 months to 12 years. Primary carers will be asked to provide informed consent whereby the children and primary carers will be enrolled into the study and followed up for 12 weeks.

DETAILED DESCRIPTION:
BACKGROUND: Malnutrition and Human Immunodeficiency Virus (HIV) infection are intimately linked and present a serious health challenge in Africa. Approximately 30-50% of children in Uganda with severe acute malnutrition (SAM) are HIV infected. Studies on nutrition as a determinant of immune response and drug metabolism in malnourished children are unknown.

GAP: Clinicians have noted that certain patients deteriorate after starting ART and nutritional supplementation despite viralogical suppression and immunological improvement with a paradoxical emergence of certain opportunistic infections, electrolyte derangement and malnutrition hence IRIS or re-feeding syndrome (RF). There is paucity of data on nutrition as a determinant of immune and pharmacological response amongst HIV infected malnourished children despite malnutrition being common.

HYPOTHESIS: Well-nourished HIV infected children ART naïve or experienced will have a better nutritional, clinical, immunological and pharmacological outcome than malnourished children ART naïve or experienced.

METHODS: A cohort design studying 75 malnourished HIV infected children on ART and RUTF comparing them to 75 well-nourished children ART naive or experienced aged between 6 months to 12 years after primary carers have provided informed consent will be enrolled into the study and followed up for 12 weeks.

IMPACT: This study will endeavor to provide appropriate information that will enhance the management of malnourished HIV infected children in the context of both ART and RUTF and their impact on immune response and drug metabolism. The study will also generate other research questions that need to be addressed in order to optimize HIV services amongst malnourished children.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected children aged 6 months to 12 years, including Well Nourished (WN), Moderately Acute Malnutrition (MAM) and Severe Acute Malnutrition (SAM) patients initiating on ART within 2 weeks, whose carer is aged ≥18 years and has provided informed consent.
* Malnourished HIV-infected children aged 6 months to 12 years stabilized on ART for at least 6 months and initiating on RUTF, whose carer is aged ≥18 years and has provided informed consent.

Exclusion Criteria:

1. Previous enrollment in a nutritional therapeutic program in the last 3 months
2. Children involved in an on-going nutrition study
3. Children who have previously received the tuberculin skin test (TST) or mantoux or purified protein derivative (PPD) in the last 3 months.
4. Children with clinically suspected or confirmed malignancy
5. Children exhibiting any specific food intolerance
6. Children who are vomiting profusely (over 3 times daily)
7. Children living outside 50 km radius from Infectious Diseases Institute at Mulago, Kampala
8. Children whose carers do not want to disclose their home address.
9. Children whose cause of malnutrition is compounded by congenital malformations, chromosomal disorders, metabolic disorders, congenital immune disorders, cerebral palsy
10. Children with a severe disability limiting the possibility of investigations
11. Children who plan to leave the catchment area in the next 6 months

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-12 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Changes in numbers of circulating immune cell population and their capacity to release cytokines | 12 weeks
  Immune response

SECONDARY OUTCOMES:
Occurrence of Immune reconstitution inflammatory syndrome (IRIS) | 12 weeks
  Episodes of Opportunistic infections - Clinical outcomes
Occurrence of re-feeding syndrome | 12 weeks
  Episodes of Opportunistic infections - Clinical outcomes
Pharmacological: Cmax | 12 weeks
  Cmax of Non-nucleotide reverse - transcriptase inhibitors (NNRTI) and Protease Inhibitors(PIs) at 0weeks, 6weeks,12weeks
Pharmacological: AUC | 12 weeks
  Area Under Curve (AUC) Time Frame: 0weeks, 6weeks, 12weeks for nevirapine and lopinvir/retonavir
Number of participants with adverse events | 12 weeks
  Pharmacological: Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Judy Orikiiriza, MMED, Principal Investigator — PhD Candidate
Locations (2):
- Uganda (2):
  - Infectious Diseases Institute, Kampala, Kampala
  - Mildmay International Centre Kampala, Kampala, Kampala